CLINICAL TRIAL: NCT04164277
Title: Using Facebook and Participatory Learning in an Intergenerational Intervention to Prevent Obesity in Head Start Preschoolers
Brief Title: FirstStep2Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Jiying Ling, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21NR017958 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-15 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Obesity; Risk Reduction Behavior; Early Intervention; Intergenerational Relations
Keywords: Obesity prevention, early childhood, intergenerational, family-based
MeSH Terms: conditions — Pediatric Obesity; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: From the eligible 13 Head Start centers with at least three classrooms in one Head Start organization, six Head Start centers will be randomly selected and assigned to the intervention (n = 3) or control (n = 3) group with usual Head Start activities. Three to five classes will be randomly selected from each selected Head Start center to be involved in the study. In each class, six caregiver-preschooler dyads will be randomly selected from the eligible participants, and total 24 caregiver-preschooler dyads will be recruited from each center, yielding a total of 144 dyads.
Who Masked: Outcomes Assessor
Masking Description: Data collectors and interviewers will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The 16-week intervention includes three components:
  1. Caregiver Component. Facebook-based program including four new habit-formation tasks/week, and 3 face-to-face or virtual caregiver meetings: MSU research staff will lead the meetings at Head Start centers (weeks 1, 8, & 16) to connect caregivers to each other, offer health information, and discuss behavioral change strategies.
  2. Caregiver-Preschooler Learning. Preschoolers, using stickers, will create two letters each week regarding a food or activity presented in the center-based program that they liked or want to try at home. Letters will be sent privately to each caregiver , and caregivers will be asked to respond to the letters.
  3. Center-based Preschooler Component. Built on previous research, preschoolers will receive weekly, age-appropriate, participatory learning co-delivered by teachers and MSU student educators.
  Interventions: Behavioral: Caregiver Component.; Behavioral: Caregiver-Preschooler Learning.; Behavioral: Center-based Preschooler Component.
- Control (No Intervention): Control group will receive usual Head Start activities during intervention period. After post-intervention data collection, each control caregiver will receive all intervention supplies and a mini program including a face-to-face or virtual caregiver meeting and 1-week preschooler program. The caregiver meeting will cover contents on alternative cooking ingredients, food labels, and portion sizes.

INTERVENTIONS:
Behavioral: Caregiver Component. — Facebook-based program including four new habit-formation tasks/week. Three face-to-face or virtual caregiver meetings: Meeting 1: Study orientation and healthy cooking education will be offered, and each family will receive a small bag of groceries to facilitate preparation of a recipe at home. Each caregiver will also receive an intervention cookbook containing affordable slow-cooking recipes, quick-fix recipes, and healthy snack ideas. Meeting 2: Study interveners will demonstrate how to spend less and shop healthy and how to read nutrition fact labels to promote healthy purchasing behaviors. Meeting 3: Study interveners will present healthy eating and PA community resources (e.g., farmer's markets, community gardens, nearly parks or other free or affordable PA facilities) and provide caregivers a resource booklet.
  Arms: Intervention
Behavioral: Caregiver-Preschooler Learning. — Preschoolers, using stickers, will create two letters each week regarding a food or activity presented in the center-based program that they liked or want to try at home. Letters will be sent by the PM privately to each caregiver via Facebook messenger on two weekdays. Caregivers will be asked to answer two Facebook multiple-choice questions related to the letters each week by Sunday midnight (e.g., what foods listed in the their child's letter did the participant provide? and what activities listed in the their child's letter did the participant's family try?). Caregiver responses to the questions will be summed to indicate caregiver responses to child requests. Each preschooler's letters will be kept in his/her intervention binder with other intervention materials to present to his/her caregiver at Meeting 3. Weekly preschooler activities, with pictures or videos, will be shared with caregivers via the Facebook private group every week.
  Arms: Intervention
Behavioral: Center-based Preschooler Component. — Built on previous research, preschoolers will receive weekly, age-appropriate, participatory learning co-delivered by teachers and MSU student educators. Session duration will be 20 minutes because children's normal attention span is 3-5 minutes per year of age, and 20 min/session is recommended for preschoolers. The already developed "Eat & Walk My ABCs" curriculum will be implemented. The curriculum includes four components: healthy eating learning, taste-testing activities, movement skill training, and fun physical activity.
  Arms: Intervention

SUMMARY:
This project will determine the preliminary efficacy of an innovative intergenerational intervention among Head Start preschoolers, aged 3-5 years, and their caregivers. A two-group cluster randomized controlled trial will be conducted. Six Head Start centers will be randomly assigned to the intervention (n=3) or control group (n=3), and an average of 6 caregiver-preschooler dyads will be recruited from each class (N=144 dyads from 16 classes). Grounded in an Actor-Partner Interdependence Model, the 16-week intervention has 3 components: 1) a caregiver component, including 1a) a Facebook-based program with weekly electronic retrievable flyers providing health information and behavioral change strategies and 4 weekly habit-formation tasks to improve parenting practices and home environment for preschoolers; and 1b) 3 face-to-face or virtual meetings (weeks 1, 8, & 16) to establish personal connections and communication networks among caregivers, discuss strategies, and share community resources to support preschoolers' behavioral changes at home; 2) a caregiver-preschooler learning component via Facebook messenger to send preschooler letters to each caregiver privately by the research team twice per week to 2a) share the preschooler's experiences of learning at school and his/her interests for a healthy diet and physical activity at home, and 2b) elicit caregivers' response to the letters; and 3) a Head Start center-based preschooler component to help preschoolers establish healthy habits via weekly healthy diet and physical activity participatory learning.

DETAILED DESCRIPTION:
The purpose of this two-group cluster randomized controlled trial is to determine the preliminary efficacy of an innovative intergenerational intervention on improving preschoolers' moderate-to-vigorous physical activity and diet quality, and decreasing screen time, proportion of overweight and obesity, and body mass index z-score among Head Start preschoolers (aged 3-5 years) and their caregivers.

The intervention is guided by an Actor-Partner Interdependence Model, and will target both individual-level factors, including knowledge, self-efficacy, and skill, and socio-environmental factors, including parental support for child, parenting practices, and the home environment. The 16-week intervention has three components: 1) a caregiver component including 1a) a Facebook-based program with weekly electronic retrievable flyers providing health information and behavioral change strategies, and four weekly habit-formation tasks to create a healthier home environment for preschoolers; and 1b) three face-to-face or virtual meetings (weeks 1, 8, & 16) to establish personal connections and communication networks among caregivers and discuss strategies and share community resources to support behavioral changes at home; 2) a caregiver-preschooler learning component via Facebook messenger to send preschooler letters to each caregiver privately by the research team twice per week to share the preschooler's experiences of learning at school and his/her stated interests for healthy diet and physical activity at home, and to ask caregivers to respond to the letters; and 3) a Head Start center-based preschooler component to help preschoolers establish healthy habits via weekly healthy diet and PA participatory learning.

From the eligible 13 Head Start centers with at least three classrooms in one Head Start organization, six Head Start centers will be randomly selected and assigned to the intervention (n = 3) or control (n = 3) group with usual Head Start activities. Three to five classes will be randomly selected from each selected Head Start center to be involved in the study. In each class, six caregiver-preschooler dyads will be randomly selected from the eligible participants, and total 24 caregiver-preschooler dyads will be recruited from each center, yielding a total of 144 dyads.

Three specific AIMS are:

AIM 1: Determine the preliminary efficacy of FirstStep2Health vs control among preschoolers on improving proximal behavioral changes of moderate to vigorous physical activity measured by accelerometry (primary outcome); diet quality (e.g., fruits/vegetables, fiber, whole grains, total protein, dairy, sugar-sweetened beverages, total sugars/fats), and screen time (e.g., watching television, playing video games); and decreasing distal anthropometric outcomes of proportion of overweight or obese and body mass index z-score. The investigators expect an overall decrease in body mass index z-score in intervention preschoolers because overweight or obese preschoolers' body mass index z-score is expected to decrease while healthy-weight preschoolers will have no change. The investigators focus on proximal behavioral changes as our primary outcome instead of distal anthropometric outcomes due to the brevity of this study and the need for behavioral changes to be maintained for at least a year before manifesting in changes in anthropometric outcomes.

AIM 2: Examine the preliminary efficacy of FirstStep2Health vs control among caregivers on increasing their moderate to vigorous physical activity measured by accelerometry and diet quality; decreasing their screen time, proportion of overweight or obese, and body mass index; and improving their knowledge, feeding practice skill, self-efficacy, parental support of their child, parenting practices, and home environment.

AIM 3: Compare FirstStep2Health vs control on the bidirectional relationship between preschoolers and caregivers on moderate to vigorous physical activity, diet quality, and screen time.

Further, the investigators will validate established feasibility, acceptability, and satisfaction of the intervention using qualitative and quantitative data.

This study forms the foundation for conducting a future large-scale randomized controlled trial to reduce overweight and obesity among low-income preschoolers and their caregivers.

ELIGIBILITY:
Inclusion Criteria. There are ten inclusion criteria (five for preschoolers and five for caregivers).

Preschoolers must:

1. Have parental consent.
2. Have child assent if the child is 5 years old.
3. Be 3-5 years of age. The investigators prioritize this age group because intervening with preschoolers before age 5 results in better short- and long-term weight reduction outcomes than with children older than 5; and children who are at least 3 years-old have the motor and cognitive development to participate in a healthy eating and physical activity curriculum.
4. Be able to understand and speak English. The intervention will be delivered in English.
5. Be enrolled in the full-day or part-day Head Start program. Head Start offers part-day and full-day programs. To increase the generalizability of the study findings, preschoolers from both full-day and part-day programs will be recruited in this study.

Caregivers must:

1. Provide consent.
2. Be the primary adult caregiver (≥ 18 years old) for the preschooler. Primary caregiver refers to the one person most responsible for providing care to the preschooler on a daily basis.
3. Be able to read, understand, and speak English. The intervention will be delivered in English.
4. Have at least weekly Internet access using a smartphone, tablet, or a computer. Each caregiver needs to have Internet access to access the study Facebook site for participating in the Facebook-based program.
5. Be willing to use Facebook. Since the caregiver intervention component will be delivered via Facebook, caregivers need to be willing to use Facebook in the study.

Exclusion Criteria. There are three exclusion criteria for both caregivers and preschoolers.

1. Preschoolers or caregivers who have medical conditions precluding participating in dietary changes or physical activity.
2. Preschoolers or caregivers who have diagnosed health conditions known to impact weight (e.g., Prader-Willi Syndrome) or are taking weight-affecting medications (e.g., stimulants).
3. Preschoolers who have diagnosed developmental disabilities (e.g., autism), or caregivers who have diagnosed psychiatric or mental health problems.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Area Community Services, Inc. Head Start and Early Childhood Programs, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other investigators upon request after securing a completed Data Use Agreement. We will adhere to the NIH Policy for Data Sharing from Clinical Trials and Epidemiological Studies. We will make any data not previously released and other study materials not previously distributed to individuals who are not study investigators available within three years of the end of NIH support for the study in accordance with the NIH Policy for Data Sharing. Only data that are stripped of personal identifiers and any personal health information will be shared.
Supporting Information: SAP, CSR
Time Frame: Within three years of the end of NIH support for the study in accordance with the NIH Policy for Data Sharing
Access Criteria: Data will be shared with other investigators upon request after securing a completed Data Use Agreement.

REFERENCES:
- [Derived] Ling J, Kao TA, Robbins LB, Kerver JM, Zhang N, Shi Y. Effects of the dyadic FirstStep2Health intervention on parents' behaviour and anthropometric outcomes: a secondary analysis of a cluster randomised trial. BMJ Open. 2024 Dec 5;14(12):e081578. doi: 10.1136/bmjopen-2023-081578. PMID 39638602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 caregiver-preschoolers dyads (53 caregivers, 53 preschoolers) from 10 daycare centers were enrolled in the study, and 10 daycare centers were randomly assigned into the intervention (5 daycare centers, 53 dyads) and control (5 daycare centers, 42 dyads) group.
Units Other Than Participants: Daycare centers
Period: Preschoolers
Arm/Group | Intervention | Control
Started (53 preschoolers in 5 intervention daycare centers and 42 preschoolers in 5 control intervention dyads) | 53; 5 Daycare centers | 42; 5 Daycare centers
Completed (47 preschoolers in 5 intervention daycare centers and 36 preschoolers in 5 control intervention dyads) | 47; 5 Daycare centers | 36; 5 Daycare centers
Not Completed | 6; 0 Daycare centers | 6; 0 Daycare centers
Period: Caregivers
Arm/Group | Intervention | Control
Started | 53; 5 Daycare centers | 42; 5 Daycare centers
Completed | 47; 5 Daycare centers | 36; 5 Daycare centers
Not Completed | 6; 0 Daycare centers | 6; 0 Daycare centers

BASELINE CHARACTERISTICS:
Population: The baseline sample included 53 caregiver-preschooler dyads (total 106 individuals, 53 caregivers, 53 preschoolers) in the intervention group and 42 caregiver-preschooler dyads (total 84 individuals, 42 caregivers, 42 preschoolers) in the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 106 | 84 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data from caregivers and preschoolers were analyzed separately.
  Years
    Preschoolers: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers | 4.12 (0.56) | 4.09 (0.57) | 4.11 (0.56)
    Caregivers: number analyzed (Participants) | 53 | 42 | 95
    Caregivers | 30.74 (6.11) | 30.02 (5.27) | 30.42 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data from caregivers and preschoolers were analyzed separately. Caregivers could select more than one choice and one caregivers selected both "female" and "male."
  Participants
    Preschoolers: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: Female | 26 | 29 | 55
    Preschoolers: Male | 27 | 13 | 40
    Caregivers: number analyzed (Participants) | 52 | 42 | 94
    Caregivers: Female | 48 | 39 | 87
    Caregivers: Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data from caregivers and preschoolers were analyzed separately. Participants could select more than one choice making the Rows not mutually exclusive.
  Participants
    Preschoolers: Hispanic preschoolers: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: Hispanic preschoolers | 7 | 5 | 12
    Preschoolers: White or Caucasian: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: White or Caucasian | 10 | 21 | 31
    Preschoolers: Black or African American: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: Black or African American | 24 | 14 | 38
    Preschoolers: Asian/Pacific Islander: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: Asian/Pacific Islander | 3 | 0 | 3
    Preschoolers: Mixed Race: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: Mixed Race | 15 | 7 | 22
    Preschoolers: American Indian or Alaskan Native: number analyzed (Participants) | 53 | 42 | 95
    Preschoolers: American Indian or Alaskan Native | 1 | 0 | 1
    Caregivers: Hispanic: number analyzed (Participants) | 53 | 42 | 95
    Caregivers: Hispanic | 3 | 5 | 8
    Caregivers: White or Caucasian: number analyzed (Participants) | 53 | 42 | 95
    Caregivers: White or Caucasian | 18 | 26 | 44
    Caregivers: Black or African American: number analyzed (Participants) | 53 | 42 | 95
    Caregivers: Black or African American | 23 | 12 | 35
    Caregivers: Asian/Pacific Islander: number analyzed (Participants) | 53 | 42 | 95
    Caregivers: Asian/Pacific Islander | 3 | 0 | 3
    Caregivers: Mixed race: number analyzed (Participants) | 53 | 42 | 95
    Caregivers: Mixed race | 6 | 3 | 9
    Caregivers: American Indian or Alaskan Native: number analyzed (Participants) | 53 | 42 | 95
    Caregivers: American Indian or Alaskan Native | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 106 | 84 | 190

OUTCOME MEASURES:

1. Primary Outcome: Moderate-to-vigorous Physical Activity (MVPA; Preschoolers)-AIM 1
Description: The ActiGraph GT3X accelerometer (www.theactigraph.com) will record acceleration counts from which minutes of MVPA per day will be estimated (analysis software available). Each caregiver-preschooler dyad will receive the accelerometers at the same time and data collectors will explain to both caregiver and preschooler how to wear the accelerometers. Preschoolers' caregivers will be instructed to return monitors either at the Head Start center or via mail using using the provided prepaid envelope after the seventh day. Data will be downloaded to the same computer used to initialize monitors. Initial analysis will use 15-sec. epochs and the following count thresholds: moderate (420-841 counts/15 seconds) and vigorous PA (≥ 842 counts/15 seconds). Fifteen-second increments with counts ≥ 420 will be summed to determine minutes of MVPA.
Time Frame: Moderate-to-vigorous physical activity at 17 weeks
Measure: Mean (Standard Deviation); unit: Minutes per hour
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Minutes per hour | 7.51 (3) | 7.46 (2.17)

2. Secondary Outcome: Fruit/Vegetable Intake (Preschoolers)-AIM 1
Description: Preschoolers' fruit/vegetable intake (servings/day) at home will be assessed by three non-consecutive 24-hour dietary recalls (one weekend day; two weekdays; randomly selected) with their caregivers over 2-3 weeks. The Project Manager will be trained at the University of Minnesota Nutrition Coordinating Center for two days and certified. The Project Manager will train interviewers to collect data individually from each caregiver via telephone. To aid in assessment of portion sizes, two-dimensional food models and measuring guides will be provided to caregivers at Head Start centers. Preschoolers' dietary intake at the Head Start center will be assessed by the dietary observation system on snacks and lunch on two selected weekdays (similar to the two weekdays selected for the 24-hour recall). The observed diet data will be entered into the Minnesota Nutrition Data System for Research for analysis.
Time Frame: Fruit/vegetable intake at 17 weeks
Measure: Mean (Standard Deviation); unit: Servings per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Servings per day | 3.60 (2.01) | 3.61 (2.68)

3. Secondary Outcome: Screen Time (Preschoolers)-AIM 1
Description: Preschoolers' screen time will be assessed by two questions from the National Health and Nutrition Examination Survey (NHANES)-Physical Activity and Physical Fitness Survey. The two questions ask caregivers about the number of hours per day their preschooler watches television or videos and uses a computer or plays games. The scale has good reliability with coefficients ranging from 0.63 to 0.84. The sum score of the two questions (min-max: 0-24 hours/day) will be used to describe preschoolers' screen time, with a higher score indicating more screen time. Caregivers will complete the survey.
Time Frame: Screen time at 17 weeks
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Hours per day | 3.70 (2.99) | 3.58 (2.71)

4. Secondary Outcome: Number of Preschoolers Who Are Overweight or Obese-AIM 1
Description: Data collectors will measure each preschooler (bulky clothing, shoes, and things in pockets removed) in a private room. In accordance with NHANES measurement protocol, height without shoes will be measured to the nearest 0.1 cm. with a Shorr Board (Weigh and Measure, LLC, Olney, MD), and weight in kg. will be measured to the nearest 0.1 kg. using a Seca model 874 portable electronic scale (Seca Corp., Columbia, MD). Two measurements will be taken for height and weight. If the two differ by < 0.5 cm. and < 0.5 kg., they will be averaged to determine the final height and weight, respectively. If the two measurements differ by ≥ 0.5 cm. or by ≥ 0.5 kg, a third one will be taken. If the 3rd measurement is ≥ 0.5 cm or ≥ 0.5 kg. different from the previous two measurements, process will be repeated and another data collector will measure. BMI percentile and BMI z-score for age and sex will be determined via SAS program for CDC Growth Charts.
Time Frame: Proportion of overweight and obesity at 17 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Participants | 14 | 12

5. Other Pre Specified Outcome: Moderate-to-vigorous Physical Activity (MVPA; Caregivers)-AIM 2
Description: The ActiGraph GT3X-plus accelerometer (www.theactigraph.com) will record acceleration counts from which minutes of MVPA per day will be estimated (analysis software available). Data collection procedure for caregivers will be similar to those employed for preschoolers, but different count thresholds will be used: moderate (2690-6166 counts/60 seconds) and vigorous PA (≥ 6167 counts/60 seconds). Sixty-second increments with counts ≥ 2690 will be summed to determine minutes of MVPA.
Time Frame: Moderate-to-vigorous physical activity at 17 weeks
Measure: Mean (Standard Deviation); unit: Minutes per hour
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Minutes per hour | 8.25 (6.75) | 10.14 (9.77)

6. Other Pre Specified Outcome: Fruit/Vegetable Intake (Caregivers)-AIM 2: Block Fruit-Vegetable-Fiber Screener
Description: The ten-item Block Fruit-Vegetable-Fiber Screener will assess the caregivers' fruit/vegetable intake (servings/day). This survey provides estimates for intake of food groups including total fruit/vegetable servings, dietary fiber (mg), Vitamin C (mg), magnesium (mg), and potassium (mg). The scale is significantly correlated with the full Block survey (r = 0.71). The established scoring equation will be used to calculate the number of servings of fruit/vegetable each participant consumes per day.
Time Frame: Diet quality at 17 weeks
Measure: Mean (Standard Deviation); unit: Servings per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Servings per day | 4.52 (2.46) | 3.44 (1.58)

7. Other Pre Specified Outcome: Screen Time (Caregivers)-AIM 2
Description: Caregivers' screen time will also be assessed by two questions from the National Health and Nutrition Examination Survey (NHANES)-Physical Activity and Physical Fitness Survey. The sum of the two questions (min-max: 0-24 hours/day) will be used to describe preschoolers' screen time, with a higher score indicating more screen time.
Time Frame: Screen time at 17 weeks
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Hours per day | 4.93 (4.71) | 5.93 (5.67)

8. Other Pre Specified Outcome: Number of Caregivers Who Are Overweight or Obese-AIM 2
Description: BMI will be calculated based on weight (kg)/height (m2) and used to determine caregivers' weight status. Data collection procedures for caregivers will be similar to those employed for preschoolers.
Time Frame: Proportion of overweight and obesity at 17 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 20
Participants | 23 | 16

9. Other Pre Specified Outcome: Knowledge (Caregivers)-AIM 2
Description: The 25-item Parental Knowledge Scale will be used to assess parental knowledge on preschoolers' dietary intake and physical activity. The 2-point Likert scale has been used with low-income parents. It has two subscales: nutrition knowledge (score range 0-10), and physical activity knowledge (score range 0-15), with a higher sum score indicating greater knowledge on healthy eating or physical activity.
Time Frame: Knowledge at 17 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
score on a scale
  Nutrition knowledge | 7.45 (1.27) | 6.68 (1.87)
  Physical activity knowledge | 12.53 (1.64) | 11.58 (8.18)

10. Other Pre Specified Outcome: Feeding Practice Skill (Caregivers)-AIM 2
Description: Parent feeding practice skill will be assessed by the 33-item Child Feeding Questionnaire. The Child Feeding Questionnaire was developed to evaluate parental beliefs, attitudes, and practices regarding child feeding, with a focus on obesity proneness in children aged 2-11 years old. The 5-point Likert questionnaire, with good reliability and validity, includes seven factors: perceived responsibility, perceived caregiver weight, perceived child weight, concerns about child weight, pressure to eat, restriction, and monitoring. The mean score of the items for each factor, with a range from 1 to 5, will be calculated, with a higher mean score indicating greater perceived responsibility, perceived caregiver weight, perceived child weight, concerns about child weight, pressure to eat, restriction, and monitoring, respectively.
Time Frame: Feeding practice skill at 17 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
score on a scale
  Feeding responsibility | 4.65 (0.71) | 4.58 (0.64)
  Perceived parent weight | 3.11 (0.43) | 3.31 (0.46)
  Perceived child weight | 2.95 (0.32) | 2.88 (0.29)
  Concern about child weight | 1.46 (1.05) | 1.13 (0.26)
  Restriction | 3.33 (0.86) | 3.37 (0.87)
  Pressure to eat | 2.86 (0.99) | 2.68 (0.80)
  Monitoring | 4.04 (1.10) | 4.13 (0.83)

11. Other Pre Specified Outcome: Self-efficacy (Caregivers)-AIM 2
Description: The 20-item Parental Self-Efficacy Scale, measuring caregivers' confidence to support their preschoolers' healthy eating and physical activity, will assess caregiver self-efficacy. The 10-point Likert scale has shown good reliability with Cronbach's alphas ranging from 0.72 to 0.94. It has two subscales: nutrition self-efficacy (12 items) and physical activity self-efficacy (8 items). The mean score, with a range from 0 to 10, will be calculated for each subscale, with a higher mean score indicating greater self-efficacy.
Time Frame: Self-efficacy at 17 weeks
Measure: Mean (Standard Deviation); unit: Mean score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Mean score
  Nutrition self-efficacy | 8.95 (1.35) | 8.18 (1.68)
  Physical activity self-efficacy | 9.27 (1.12) | 8.38 (1.70)

12. Other Pre Specified Outcome: Parental Support (Caregivers)-AIM 2
Description: The 12-item Parental Support Scale for Eating Habits and Physical Activity will measure support for the child. The 6-point Likert scale has very good reliability with Cronbach's alphas ranging from 0.83 to 0.87. It has two subscales: nutrition support (7 items) and physical activity support (5 items). The mean score, with a range from 1 to 6, will be calculated for each subscale, with a higher mean score indicating greater parental support.
Time Frame: Parental support at 17 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
score on a scale
  Nutrition support | 4.52 (0.80) | 4.39 (0.71)
  Physical activity support | 5.15 (1.05) | 4.64 (1.25)

13. Other Pre Specified Outcome: Parenting Practices (Caregivers)-AIM 2
Description: The 32-item Parenting Style and Dimensions Questionnaire will measure parenting practices. The 5-point Likert questionnaire is assessing three parenting styles: authoritative, authoritarian, and permissive. The questionnaire has good reliability with Cronbach's alphas ranging from 0.64 to 0.91. The mean score of items for each parenting style, with a range from 1 to 5, will be calculated, with a higher mean score indicating greater authoritative, authoritarian, or permissive parenting style, respectively.
Time Frame: Parenting practices at 17 weeks
Measure: Mean (Standard Deviation); unit: Mean score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
Mean score
  Authoritative | 4.35 (0.52) | 4 (0.76)
  Authoritarian | 2.46 (1.24) | 2.78 (0.91)
  Permissive | 2.16 (0.84) | 2.41 (0.88)

14. Other Pre Specified Outcome: Home Environment (Caregivers)-AIM 2
Description: The 20-item Family Nutrition and Physical Activity (FNPA) screening tool will assess the home environment. This 4-point Likert screening tool is used to assess home obesogenic environments and practices, including family meals, family eating practices, food choices, beverage choices, restriction/reward, screen time, healthy environment, family activity, child activity, and family schedule/sleep routine. It has two subscales: eating environment (10 items) and physical activity environment (10 items). The sum score of the 10 items, with a range from 20 to 40, will be calculated for each subscale, with a higher sum score indicating a healthier home environment.
Time Frame: Home environment at 17 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 42
score on a scale
  Eating environment | 31.68 (4.13) | 30.74 (4.07)
  Physical activity environment | 31.24 (4.78) | 28.42 (4.71)

ADVERSE EVENTS:
Time Frame: Two years
Description: The study participants are general preschoolers and their caregivers with relatively good health, so all-cause mortality rate is expected to be 0 among the 95 participants based on the rate of 1,043.8 deaths per 100,000 population in the US.
Groups:
- Intervention - Preschoolers; Intervention - Caregivers: The 16-week intervention includes three components:
  1. Caregiver Component. Facebook-based program including four new habit-formation tasks/week, and 3 face-to-face or virtual caregiver meetings: MSU research staff will lead the meetings at Head Start centers (weeks 1, 8, & 16) to connect caregivers to each other, offer health information, and discuss behavioral change strategies.
  2. Caregiver-Preschooler Learning. Preschoolers, using stickers, will create two letters each week regarding a food or activity presented in the center-based program that they liked or want to try at home. Letters will be sent privately to each caregiver , and caregivers will be asked to respond to the letters.
  3. Center-based Preschooler Component. Built on previous research, preschoolers will receive weekly, age-appropriate, participatory learning co-delivered by teachers and MSU student educators.
- Control - Preschoolers; Control - Caregivers: Control group will receive usual Head Start activities during intervention period. After post-intervention data collection, each control caregiver will receive all intervention supplies and a mini program including a face-to-face or virtual caregiver meeting and 1-week preschooler program. The caregiver meeting will cover contents on alternative cooking ingredients, food labels, and portion sizes.
Arm/Group | Intervention - Preschoolers | Control - Preschoolers | Intervention - Caregivers | Control - Caregivers
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/42 | 0/53 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/42 | 0/53 | 0/42
Other Adverse Events (participants affected / at risk) | 0/53 | 0/42 | 0/53 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT04164277/Prot_SAP_000.pdf